CLINICAL TRIAL: NCT05399784
Title: Postpartum Visit Timing and the Effect on Visit Attendance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Kole_ConstanceHowesGrant_2020
Record Dates: First submitted 2021-10-20; First posted 2022-06-01 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Postpartum Disorder; Postpartum Depression; Postpartum Weight Retention; Breastfeeding; Satisfaction, Patient; Trust
MeSH Terms: conditions — Puerperal Disorders; Depression, Postpartum; Gestational Weight Gain; Breast Feeding; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early & Often Postpartum Care (Experimental): Visit at 2-3 and 6 weeks postpartum.
  Interventions: Behavioral: Early postpartum visit; Behavioral: Standard postpartum visit
- Standard Postpartum Care (Placebo Comparator): Visit at 6 weeks postpartum.
  Interventions: Behavioral: Standard postpartum visit

INTERVENTIONS:
Behavioral: Early postpartum visit — The early postpartum visit will be an in-person visit with a medical provider at 14-21 days postpartum.
  Arms: Early & Often Postpartum Care
Behavioral: Standard postpartum visit — The standard postpartum visit will occur at 35 to 56 days postpartum.

SUMMARY:
The objective of this study is to assess if the addition of an early postpartum visit improves attendance at postpartum visits. We seek to evaluate if an additional early postpartum visit improves patient education, satisfaction, or trust in the clinicians during the postpartum period; all of which may ultimately facilitate improved outcomes. Additionally, we seek to explore patient preferences for postpartum care delivery.

DETAILED DESCRIPTION:
Maternal mortality in the United States is currently at a record high of 17 deaths per 100,000 live births and the majority of pregnancy related deaths occur in the postpartum period due to complications from chronic disease exacerbation, pregnancy-related hypertension, or psychiatric conditions that lead to suicide. Optimal postpartum care would reduce mortality risk, but numerous studies have demonstrated current care is inadequate. Up to 40% of women do not attend their postpartum visit at 4-6 weeks after delivery and the 15-minute visit is too short to achieve the comprehensive goals that the American College of Obstetricians and Gynecologists (ACOG) sets for this visit: a full assessment of physical, social, and psychological well-being. In addressing the current gap between optimal and actual care, ACOG recently recommended that practitioners shift from the standard, single six-week postpartum visit to two postpartum visits, the first within three weeks of delivery. While this change is intended to address current sub-optimal outcomes, the effects of this change are entirely unknown.

The long term goal of our program is to improve postpartum care for women in Rhode Island. The primary objective of this project is to determine if the ACOG proposed additional postpartum visit within three weeks of delivery improves attendance to postpartum appointments compared to routine postpartum care. Additionally, we intend to examine whether having two scheduled postpartum visits (one within three weeks and the other at the standard 4-6 week postpartum time point) which we describe as "early and often" postpartum care-improves patient knowledge, satisfaction and trust in clinicians compared to routine care as well as explore patient preferences for postpartum care. Our central hypothesis is that early and often postpartum care will lead to improved patient visit attendance compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

* age 13 to 50 years old
* literacy in English or Spanish
* receipt of prenatal care at the Obstetrics and Gynecology Care Center of Women & Infants Hospital
* delivery at Women & Infants Hospital during the study time period

Exclusion Criteria:

High risk pregnancy defined as one or more of the following:

* chronic hypertension
* gestational hypertension
* preeclampsia
* eclampsia
* third degree perineal laceration
* fourth degree perineal laceration
* blood product transfusion
* intensive care unit admission
* who were prescribed anxiolytic or antidepressant medications in the antepartum period

Ages: 13 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 162 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Number of postpartum visits attended | 3 months
  The number of times a patient attends a postpartum visit in the first 12 weeks postpartum will be counted

SECONDARY OUTCOMES:
Number of recommended items covered during postpartum care | 3 months
  Patients will complete a survey (created for this study) and identify how many key postpartum items were discussed during their postpartum care.
Trust in physician scale | 3 months
  The Trust in Physicians scale is a reliable and valid measure of a patients trust in their clinician and has been shown to be distinct from patient satisfaction
Short Assessment of Patient Satisfaction | 3 months
  The Short Assessment of Patient Satisfaction (SAPS) is a short, reliable, valid, seven item scale to assess patients satisfaction with medical treatment and care
Number of emergency room visits | 3 months
  Emergency room utilization will be determined via the electronic medical record. The number of visits in the first 3 months postpartum will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Martha B Kole-White, MD, Principal Investigator — Women & Infants Hospital
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No